CLINICAL TRIAL: NCT06113380
Title: Effect on Upper Limb Training Using Rehabilitation Robot With Human-Computer Interaction Game Interface for Stroke Patients
Brief Title: Using Upper Limb Rehabilitation Robot in Stroke Patient Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201905073DINC
Record Dates: First submitted 2023-10-25; First posted 2023-11-02 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation by rehabilitation robot (Experimental): Rehabilitation therapists will determine the training mode based on the subject's movement ability.
  Passive training mode Active-assistive training mode
  Interventions: Device: NTUH-ii, am upper limb rehabilitation robot arm
- Traditional rehabilitation (Active Comparator): Traditional upper limb physical therapy is performed by the therapist.
  Interventions: Other: Traditional upper limb physical therapy

INTERVENTIONS:
Device: NTUH-ii, am upper limb rehabilitation robot arm — Rehabilitation programs are planned based on the subject's capabilities, and the differences between assisted rehabilitation with a robot and traditional rehabilitation are compared.
  Arms: Rehabilitation by rehabilitation robot
Other: Traditional upper limb physical therapy — Traditional upper limb physical therapy is performed by the therapist.
  Arms: Traditional rehabilitation

SUMMARY:
A robot arm for upper limb rehabilitation is intended to achieve rehabilitation effects through the study of robot control theory and the integration of sensors such as sEMG. The goal is to reduce the workload of rehabilitation therapists.

DETAILED DESCRIPTION:
NTUH-ii is an upper limb rehabilitation robot. The aim of this robot is to reduce the workload of rehabilitation therapists and make the rehabilitation process more effective.

The robot can complete rehabilitation tasks, such as elbow flexion/extension, shoulder flexion/extension, and shoulder horizontal abduction/adduction, etc. By giving the desired trajectory, the robot can lead patients to do the tasks in passive mode or active mode.

However, curative rehabilitation should include the motion intention of patients. This study aimed to investigate the efficacy of rehabilitation effect by combining the sensors (such as sEMG, IMU) to obtain the motion intention of patients and give the assistive movement.

ELIGIBILITY:
Inclusion Criteria:

1. First-time stroke, occurring between 2 weeks and 2 years after onset, resulting in unilateral hemiplegia.
2. Able to understand and follow simple instructions.
3. Able to maintain a sitting posture balance.
4. Rank on the Brunnstrom Scale is between two and five.
5. Both ischemic and hemorrhagic strokes are included.

Exclusion Criteria:

1. Not yet fully conscious.
2. Suffering from a psychiatric disorder or post-stroke psychiatric abnormalities.
3. Cognitive or behavioral impairments that affect the ability to comprehend or execute the experimental tasks.
4. Severe aphasia preventing compliance with researchers' instructions for this study.
5. Medical conditions in internal medicine that jeopardize patient safety, such as severe heart or lung diseases, or patients requiring bed rest.
6. Patients with a severe systemic illness requiring bed rest.
7. Patients with shoulder joint pathology unable to undergo exercise therapy.
8. Patients with severe osteoporosis who have concerns about fractures during physical activity.
9. Patients with arrhythmia and implanted cardiac pacemakers.
10. Severe uncontrolled seizures that cannot be improved with medication, physical therapy, botulinum toxin injections, or phenol block procedures.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment | 1 month
  Fugl-Meyer assessment upper extremity, higher scores indicate a better outcome.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment | Before the task and right away the experiment, 3 months, 6 months post intervention.
  Fugl-Meyer assessment upper extremity, higher scores indicate a better outcome.
sEMG analyzation | Before the task, right away the experiment and 1 month, 3 months, 6 months post intervention.
  using sEMG sensors to obtain the sEMG signal and applying 3×2 ANOVA to analyze.
Modified Ashworth Scale | Before the task, right away the experiment and 1 month, 3 months, 6 months post intervention.
  To measure the increase of muscle tone, score from 0 to 4, higher scores indicate the higher muscle tone.
Wolf Motor Function Test | Before the task, right away the experiment and 1 month, 3 months, 6 months post intervention.
  To quantify upper extremity movement ability through timed single- or multiple-joint motions .and functional tasks.
Stroke Impact Scale | Before the task, right away the experiment and 1 month, 3 months, 6 months post intervention.
  A self-report questionnaire that evaluates disability and health-related quality of life after stroke. Score from 0 to 100, Higher scores indicate a better outcome.
Motor evoked potential | Before the task, right away the experiment and 1 month, 3 months, 6 months post intervention.
  action potential elicited by noninvasive stimulation of the motor cortex

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No